CLINICAL TRIAL: NCT04926090
Title: Developing Supports to Address Mental Health Needs of Autistic Students in Postsecondary Education
Brief Title: Developing Mental Health Supports for Autistic Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Principal Investigator, Vanessa H. Bal, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2021000076
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder; Depression, Anxiety
Keywords: smartphone; ecological momentary intervention (EMI); ecological momentary assessment (EMA)
MeSH Terms: conditions — Autism Spectrum Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional Support Plan - Clinician Guided (ESP-C) + (Bi)Weekly Monitoring (Experimental): This will involve brief assessment visits throughout the fall semester, without prompting to use the ESP-C. Visits will be weekly for the first 6 weeks and then biweekly for the remaining 9 weeks of the term.
  Interventions: Behavioral: Emotional Support Plan - Clinician Guided (ESP-C)
- Emotional Support Plan - Clinician Guided (ESP-C) + 4x Daily Monitoring (Experimental): Participants in this arm will be prompted on their phones 4x/day, to report on activities, mood, suicidal ideation, distress level and ESP use since the last prompt. They will also participate in brief assessment visits conducted weekly for the first 6 weeks and then biweekly for the remaining 9 weeks of the term.
  Interventions: Behavioral: Emotional Support Plan - Clinician Guided (ESP-C)
- Emotional Support Plan - Self Guided (ESP-S) + 4x Daily Monitoring (Experimental): Participants in this arm will be prompted on their phones 4x/day, to report on activities, mood, suicidal ideation, distress level and ESP use since the last prompt. They will be asked to complete questionnaires weekly for the first 6 weeks and then biweekly for the remaining 9 weeks of the term.
  Interventions: Behavioral: Emotional Support Plan - Self Guided (ESP-S)

INTERVENTIONS:
Behavioral: Emotional Support Plan - Clinician Guided (ESP-C) — The Emotional Support Plan (ESP) is designed to help prepare students to cope with stress experienced during postsecondary education. The ESP-C is delivered by a clinician in 2 sessions.
  Arms: Emotional Support Plan - Clinician Guided (ESP-C) + (Bi)Weekly Monitoring; Emotional Support Plan - Clinician Guided (ESP-C) + 4x Daily Monitoring
Behavioral: Emotional Support Plan - Self Guided (ESP-S) — The Emotional Support Plan (ESP) is designed to help prepare students to cope with stress experienced during postsecondary education. The ESP-S is created by the participant on their own, with the support of self-guided materials.
  Arms: Emotional Support Plan - Self Guided (ESP-S) + 4x Daily Monitoring

SUMMARY:
The present study aims to expand the availability of emotional supports in order to promote successful transitions and longer-term outcomes for autistic students in PSE.

DETAILED DESCRIPTION:
This study has three specific aims:

Aim 1: Identify mental health needs of autistic students to inform supports. Focus groups engaging key stakeholders will be used to understand the mental health needs of autistic college students and inform adaptation of two individualized mental health supports: 1) the ESP intervention and 2) protocols for monitoring mood and psychological distress.

Aim 2: Develop resources to inform and guide mental health care of autistic students. Focus group information will inform 1) adaptation of clinician (ESP-C) and self-guided (ESP-S) emotional support plans and monitoring protocols and 2) develop a "College Student Mental Health Guide" to aide autistic college students, their families and mental health professionals in proactive planning for mental health supports during PSE.

Aim 3: Assess the feasibility, acceptability and initial efficacy of the ESP-C and ESP-S.

The study will yield preliminary data to apply for additional funding to conduct a large-scale trial to validate these methods to monitor and support mental health of autistic adults. Information gathered from the study will also be used to inform development of a mental health guide for autistic students.

ELIGIBILITY:
Inclusion Criteria:

* Previous ASD diagnosis,
* Has smartphone (to access the ESP app)
* At least 6th grade Reading Comprehension on the WRAT-5. The WRAT-5 may not be required if a student has other evidence of age-appropriate reading level.
* Be currently enrolled in a Postsecondary Education (PSE) institution.

Exclusion Criteria:

* Not a students in a PSE Institution or do not have diagnosis of ASD
* Score below a 6th grade Reading Comprehension on the WRAT-5
* Unable to understand English
* No access to a compatible iOS and Android smartphone
* the PI's clinical judgment that it would not be in the adult's best interest to be enrolled

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Change in distress on Patient Health Questionnaire (PHQ-9) | 15 week monitoring period
  The PHQ-9, assessed weekly for first 6 weeks and biweekly for remaining 9 weeks, is a 9-item questionnaire of psychological function over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Higher scores equal more distress.
Change in distress on Ecological Momentary Assessment (EMA) reports | 15 week monitoring period
  EMA (Ecological Momentary Assessment) reports of decreased distress (in ESP + daily monitoring groups only). Scores range from 0(not at all) to 5 (very much). Higher scores on the item equal higher levels of distress.
Change in anxiety symptoms on the Generalized Anxiety Disorder Questionnaire (GAD-7) | 15 week monitoring period
  The GAD-7, assessed weekly, is a 7-item questionnaire of anxiety symptoms over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Higher scores equal more anxiety.

SECONDARY OUTCOMES:
Change in Adult Self Report | 15 week monitoring period
  The ASR is a measure of adaptive functioning and psychopathology (e.g., anxiety, depression symptoms). Most of the items are on a 3 point scale including: (0) Not true, (1) Somewhat or sometimes true, and (2) Very often or often true. Higher scores equal more symptoms.
Change in Adult Behavior Checklist | 15 week monitoring period
  The ABCL is a caregiver-report measure of adaptive functioning and psychopathology (e.g., anxiety, depression symptoms). Most of the items are on a 3 point scale including: (0) Not true, (1) Somewhat or sometimes true, and (2) Very often or often true. Higher scores equal more symptoms.
Change in Emotion Dysregulation Inventory | 15 week monitoring period
  The EDI is a measure of emotion dysregulation designed for use with individuals with autism. Items are rated on a scale of 0-5. Higher score equal more symptoms.
Change Young Adult Coping Orientation for Problem Experience (YA-COPE) | 15 week monitoring period
  The YA-COPE is a 56-item measure designed to capture coping behaviors of college students. Items are rated on a scale of 1(never) to 5 (most of the time. Higher scores indicate more positive strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa H Bal, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No